CLINICAL TRIAL: NCT04377607
Title: An Important Index on Severity of Coronavirus Disease: Erythrocyte Haemoglobin Concentration
Brief Title: Haemoglobin Concentration on COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nevsehir Public Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif Yazar, Specialist, Nevsehir Public Hospital
Other Study IDs: 145/2020
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Corona Virus Infection
Keywords: coronavirus; haemoglobin concentration; COVID-19; severity of disease
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group OP: outpatients with asymptomatic or uncomplicated or mild pneumonia
  Interventions: Other: File scanning
- Group H: hospitalized patients
  Interventions: Other: File scanning
- Group IC: patients admitted to intensive care unit
  Interventions: Other: File scanning

INTERVENTIONS:
Other: File scanning — RBC, HGB, HCT, MCH, MCV, MCHC, WBC values will be noted in the hemogram test performed at the time of initial admission

SUMMARY:
A rapid oxygen desaturation has observed in patients with COVID-19 which have seriously respiratory failure and most of them have intubated and connected to the mechanical ventilator. Finally, many of them have died during the process.

ORF8 and superficial glycoproteins of a novel coronavirus bind to porphyrin on haemoglobin molecules and inhibit heme metabolism in an erythrocyte. However, it is not clarify the effects of the novel coronavirus on mean corpuscular volume (MCV), mean corpuscular of haemoglobin (MCH) and mean corpuscular haemoglobin concentration (MCHC).

DETAILED DESCRIPTION:
In late December 2019, cases of pneumonia of unknown etiology began to appear in Wuhan, Hubei, China. This disease, which was named COVID-19 by the World Health Organization (WHO) on February 11, 2020, was identified as serious acute respiratory syndrome coronavirus-2 (SARS-CoV-2). The disease, which spread rapidly from person to person, quickly became a pandemic in the world.

Some of the patients who admitted with high fever, cough and respiratory distress have been curing in intensive care units due to severe respiratory failure. A rapid oxygen desaturation has observed in these patients, and most of the patients have intubated and connected to the mechanical ventilator, but many of them have died in this process. Until May 02, 2020, approximately 3,5 million COVID-19 cases were detected throughout the world and nearly 250 thousand people died.

In this process, to identfy the reasons of the respiratory failure and oxygen desaturation has a high scientific value. Alveolar edema and reactive pneumocyte hyperplasia accompanied by inflammatory infiltration in the lung during the early stage of infection may cause disruption of oxygen transport. In some cases, the alveolar exudate organization and pulmonary interstitial fibrosis accompany this process, and the desquamation of the mucosal epithelium and the bronchi are covered with a mucous plug. The resulting destruction is thought to cause desaturation by affecting oxygen transport.

A novel coronavirus has a positive stranded RNA nucleic acid. In addition to its structural spikes, envelope and membrane proteins, it has non-structural proteins such as ORF1ab, ORF3a, ORF6, ORF7a, ORF10 and ORF8. Inhibitory effects of these proteins on haemoglobin may be a reason for rapid desaturation. By binding to the porphyrin of ORF8 and superficial glycoproteins on the hemoglobin, it inhibits the "heme" metabolism and patients' haemoglobin levels may be low. However, it is not clear the effects of the disease on mean corpuscular volume (MCV), mean corpuscular of haemoglobin (MCH) and mean corpuscular haemoglobin concentration (MCHC). Demonstrating the relationship between these parameters and the severity of the disease is of great importance in the treatment of the disease in terms of further studies.

The aim of this study is to reveal the effects of the disease on erythrocyte indices and to show the effectiveness of erythrocyte indices in predicting the severity of the disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients with COVID-19 test (+) using the PCR technique

Exclusion Criteria:

* Those receiving blood products or any drugs that will affect their blood values before admission
* Those patient with any hematologic diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who applied to the hospital for a coronavirus disease symptom and whose covid-19 test was positive
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2020-11-20 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Relationship between severity of disease and values of erythrocyte indices | 5 days
  The severity of disease can decrease haemoglobin concentration and destroy oxygen transport.

SECONDARY OUTCOMES:
Sensitivity of haemoglobin concentration on severity of the disease | 5 days
  Detecting of cut-off value of haemoglobine indices can predict severity of the disease

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided